CLINICAL TRIAL: NCT03518086
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel, Placebo-Controlled Induction Study of Mirikizumab in Conventional-Failed and Biologic-Failed Patients With Moderately to Severely Active Ulcerative Colitis (LUCENT 1)
Brief Title: An Induction Study of Mirikizumab in Participants With Moderately to Severely Active Ulcerative Colitis (LUCENT 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16591; I6T-MC-AMAN (Other: Eli Lilly and Company); 2017-003229-14 (EudraCT Number)
Record Dates: First submitted 2018-05-04; First posted 2018-05-08 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis
Keywords: Interleukin-23 (IL-23) antibody; IL-23p19
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Intravenous (IV) Every 4 Weeks (Q4W) (Placebo Comparator): Placebo given as an IV infusion Q4W on Weeks 0, 4, 8 for 12 weeks.
  Interventions: Drug: Placebo
- 300 Milligram (mg) Mirikizumab IV Q4W (Experimental): 300 mg mirikizumab given as an IV infusion Q4W on Weeks 0, 4, 8 for 12 weeks.
  Interventions: Drug: Mirikizumab
- Placebo IV Q4W Maximum Extended Enrollment (ME2) (Placebo Comparator): Placebo given as an IV infusion Q4W on Weeks 0, 4, 8 for 12 weeks.
  Interventions: Drug: Placebo
- 300 mg Mirikizumab IV Q4W ME2 (Experimental): 300 mg mirikizumab given as an IV infusion Q4W on Weeks 0, 4, 8 for 12 weeks.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered IV
  Other Names: LY3074828
  Arms: 300 Milligram (mg) Mirikizumab IV Q4W; 300 mg Mirikizumab IV Q4W ME2
Drug: Placebo — Administered IV
  Arms: Placebo IV Q4W Maximum Extended Enrollment (ME2); Placebo Intravenous (IV) Every 4 Weeks (Q4W)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Mirikizumab in participants with moderately to severely active ulcerative colitis (UC) who have had an inadequate response to, loss of response, or intolerant to conventional or biologic therapy for UC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC for at least 3 months prior to baseline.
* Confirmed diagnosis of moderately or severely active UC, as assessed by the modified Mayo score (MMS).
* Demonstrated an inadequate response to, a loss of response to, or an intolerance to conventional or to biologic therapy for UC.
* If female, must meet the contraception requirements.

Exclusion Criteria:

* Participants with a current diagnosis of Crohn's disease or inflammatory bowel disease-unclassified (indeterminate colitis).
* Participants with a previous colectomy.
* Participants with current evidence of toxic megacolon.
* Prior exposure to anti-IL12p40 antibodies (e.g. ustekinumab) or anti-IL-23p19 antibodies (e.g. risankizumab, brazikumab, guselkumab or tildrakizumab).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1281 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (500):
- United States (98):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Dcr-Pi, Pc, Litchfield Park, Arizona
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Physicians Research Group, Tempe, Arizona
  - Yuma Gastro LLC, Yuma, Arizona
  - Valley Gastroenterology, Arcadia, California
  - Care Access Research, Berkeley, California
  - Citrus Valley Health Partners, Covina, California
  - Valley View Internal Medicine, Garden Grove, California
  - Om Research, LLC, Lancaster, California
  - Catalina Research Institute, LLC, Montclair, California
  - California Medical Research Associates, Northridge, California
  - Gastroenterology Associates, Pasadena, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Delta Waves Sleep Disorders and Research Center, Colorado Springs, Colorado
  - Gastroenterology Consultants of Clearwater, Clearwater, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Pioneer Clinical Research, Coral Springs, Florida
  - Direct Helpers Medical Center, Hialeah, Florida
  - The Center for Gastrointestinal Disorders, Hollywood, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - SIH Research, LLC, Kissimmee, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - IMIC, Inc., Miami, Florida
  - Inpatient Research Clinic, LLC, Miami Lakes, Florida
  - Life Medical Center & Research, Inc, Miami Lakes, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Pharma Research International, Inc., Naples, Florida
  - Center for Interventional Endoscopy, Orlando, Florida
  - Clintheory Healthcare, Orlando, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Florida Digestive Specialist, St. Petersburg, Florida
  - Florida Medical Clinic LLC, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Gastrointestinal Diseases Research, Columbus, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - NorthShore University HealthSystem, Evanston, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Delta Research Partners LLC, Monroe, Louisiana
  - Tulane Univ School of Med, New Orleans, Louisiana
  - Nola Research Works, LLC, New Orleans, Louisiana
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - MNGI Digestive Health - Plymouth Endoscopy Center & Clinic, Plymouth, Minnesota
  - Care Access Research LLC, Jackson, Mississippi
  - Digestive Health Specialists, Tupelo, Mississippi
  - Washington University Medical School, St Louis, Missouri
  - Capital Health Medical Center Hopewell, Pennington, New Jersey
  - Northwell Health, Great Neck, New York
  - NYU Langone Long Island Clinical Research Associates, Lake Success, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Digestive Diseases and Endoscopy Center, Greenville, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Trinity Health Center Medical Arts, Minot, North Dakota
  - META Medical Research Institute, LLC, Dayton, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Care Access Research - Youngstown, Poland, Ohio
  - Great Lakes Medical Research, LLC, Westlake, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Digestive Disease Associates, Wyomissing, Pennsylvania
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Invocare Clinical Research Center, Mauldin, South Carolina
  - Invocare Clinical Research Center, West Columbia, South Carolina
  - Midwest Medical Care, Sioux Falls, South Dakota
  - Gastro One, Germantown, Tennessee
  - Galen Medical Group, Hixson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Digestive Health Associates of Texas, Garland, Texas
  - Houston Methodist Research Ins, Houston, Texas
  - Biopharma Informatic, Inc., Houston, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - GI and Liver Research, LLC, Webster, Texas
  - Care Access Research LLC - Salt Lake City, Ogden, Utah
  - Care Access Research LLC - Salt Lake City, Salt Lake City, Utah
  - Emeritas Research Group, Leesburg, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - The Gastroenterology Group, P.C., Reston, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
  - Allegiance Research Specialists, LLC, Milwaukee, Wisconsin
- Argentina (8):
  - Centro de Investigaciones Metabólicas (CINME), CABA, Buenos Aires
  - Mautalen Salud e Investigacion-Centro de Osteopatías Médicas, Ciudad Autonoma de Buenos Air, Buenos Aires
  - CER Instituto Medico, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Fundación de Estudios Clínicos, Rosario, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - C.I.C.E. 9 de Julio, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Centro Medico de Cordoba SA, Córdoba
- Australia (10):
  - Princess Alexandra Hospital, Harlow, Essex
  - John Hunter Hospital, Newcastle, New South Wales
  - Coastal Digestive Health, Maroochydore, Queensland
  - Mater University Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital Outpatients, Box Hill, Victoria
  - Melbourne Gastrointestinal Investigation Unit (MGIU), Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Northern Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Austria (4):
  - Krankenhaus der Barmherzigen Schwestern Wien, Vienna, Vienna
  - Medizinische Universität Innsbruck, Innsbruck
  - Universitätsklinikum Salzburg, Salzburg
  - Medical University of Vienna, Vienna
- Belgium (5):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Centre Hospitalier de Wallonie Picarde - Site Notre Dame, Tournai, Wallonne, Région
  - AZ Klina, Brasschaat
  - AZ Groeninge, Kortrijk
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (9):
  - Gastroenterology and internal medicine research institute, Edmonton, Alberta
  - The Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - GI Research Institute, Vancouver, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - Victoria Hospital, London, Ontario
  - University of Western Ontario, London, Ontario
  - Centre de santé et de services sociaux Champlain-Charles-Le Moyne, Greenfield Park, Quebec
  - Hopital Maisonneure-Rosemount, Montreal, Quebec
  - Inflammatory Bowel Disease Centre Montreal General Hospital - MUHC, Montreal, Quebec
- China (43):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, HefeiCity, Anhui
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Xiangya Hospital Central South University, Kaifu District, Changsha City
  - The Affiliated 2nd Hosp. of Third Military Med. Univ. of PLA, Chongqing, Chongqing Municipality
  - The First Hospital Affiliated to AMU (Southwest Hospital), Chongqing, Chongqing Municipality
  - Fujian Province Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Of Fujian Medical University, Fujian, Fuzhou
  - The Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - ZhuZhou Central Hospital, Zhuzhou, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Central General Hospital, Jilin, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Lianing
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital Affliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - No.1 Hospital Affiliated to Xinjiang Medical University, Ürümqi, Urumchi
  - Kunming Medical College Affiliated First Hospital, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Med, Hangzhou, Zhejiang
  - First Affiliated Hosp of College of Med, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital YuYing Childens Hospital of Wenzhou Medical university, Wenzhou, Zhejiang
  - Tongji Hospital of Tongji University, Wuhan
- Croatia (3):
  - University Hospital Center Osijek, Osijek
  - CHC Zagreb, Zagreb
  - Polyclinic Bonifarm, Zagreb
- Czechia (10):
  - Vojenska nemocnice Brno, Brno, Brno-město
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Hl. M. Praha
  - Hepato-gastroenterologie HK, Hradec Králové, Hradec Králové
  - Klinika ResTrial, Prague, Modrany
  - MUDr. Gregar, s.r.o., Olomouc, Olomoucký kraj
  - A-Shine, Pilsen, Plzeň-město
  - Mediendo, Prague, Praha 8
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - PreventaMed, s.r.o., Olomouc
  - ISCARE Clinical Centre, Prague
- Denmark (3):
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Herlev and Gentofte Hospital, Herlev
  - Zealand University Hospital Køge, Køge
- France (16):
  - Hopital de Hautepierre - Service d'Hépatogastroentérolgie, Strasbourg, Bas Rhin
  - Hopital Saint-Louis, Paris, Cedex 10
  - CHU Lille - Hôpital Claude Huriez, Lille, Nord
  - Hopital Beaujon, Clichy, Paris
  - Centre Hospitalier de Pau, Pau, Pyrénées-Atlantiques
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud -, Pierre-Bénite, Rhone
  - CHU Amiens Picardie-Site Sud - RDC Service Hépato gastro, Amiens, Somme
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Hopital Saint Eloi, Montpellier
  - Hopital L'Archet 2, Nice
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - CHU de Poitiers- Service d'Hépato-gastro-entérologie,, Poitiers
  - Robert Debre Hospital, Reims
  - CHU de Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHRU Nancy Brabois - Hôpital d'Enfants, Vandœuvre-lès-Nancy
- Germany (11):
  - Medizinische Hochschule Hanover, Hanover, Lower Saxony
  - Gastro Campus Research GbR, Münster, North Rhine-Westphalia
  - Haus der Gesundheit, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle, Saxony-Anhalt
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Charité Campus Virchow-Klinikum, Berlin
  - Krankenhaus Waldfriede, Berlin
  - Staedisches Klinikum Brandenburg, Brandenburg
  - HaFCED - Hamburgisches Forschungsinstitut für chronisch entzündliche Darmerkrankungen, Hamburg
  - Praxiszentrum Alte Maelzerei, Regensburg
  - Internistische Praxisgemeinschaft, Weyhe
- Hungary (9):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred, EU
  - Jávorszky Ödön Kórház, Vác, Pest County
  - Óbudai Egészségügyi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Endomedix Diagnosztikai Központ - Miskolc, Miskolc
  - Karolina Korhaz-Rendelointezet, Mosonmagyaróvár
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont I. Belgyogyaszati Klinika, Szeged
  - Clinfan Szolgaltato Kft., Szekszárd
- India (22):
  - Centre for Liver Research & Diagnostics, Deccan College of Medical Sciences, Owaisi Hospital & Research Centre, Hyderabad, Andhra Pradesh
  - Institute of Digestive and Liver Diseases, Guwahati, Assam
  - Apollo Research and Innovations, Apollo Hospitals International Ltd, Gandhinagar, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Nirmal Hospital, Surat, Gujarat
  - Bangalore Medical College and Research Institute, Bangalore, Karnataka
  - M S Ramaiah Medical College Hospital, Bangalore, Karnataka
  - Lokmanya Hospital, Mumbai, Maharashtra
  - Midas Multispecilaity Hopsital Pvt Ltd, Nagpur, Maharashtra
  - Poona Medical Foundation. Ruby Hall Clinic, Pune, Maharashtra
  - K E M Hospital and Research Centre, Pune, Maharashtra
  - Datta Meghe Institute of Medical Sciences (DU), Acharya Vinoba Bhave Rural Hospital, Wardha, Maharashtra
  - Escorts Heart Institute and Research Centre Ltd, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Asian Institute of Gastroenterology, Hyderabad, Telangana
  - King George Medical University, Lucknow, Uttar Pradesh
  - Fortis Hospital, Noida, Uttar Pradesh
  - SSKM Post Graduate Hospital, Kolkata, West Bengal
  - Nil Ratan Sircar Medical College, Kolkata, West Bengal
  - Gandhi Hospital, Telangana
- Beaumont Hospital, Dublin, Dublin, Ireland
- Israel (8):
  - Meir Medical Center, Kfar Saba, Central District
  - Shaare Zedek Medical Center, Bait Vagan, Jerusalem
  - Soroka Medical Center - Pediatric Outpatient Clinic, Beersheba
  - Galilee Medical Center Department of Internal Medicine A, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - King Fahad Medical City, Ẕerifin
- Italy (16):
  - Presidio di Rho, Rho, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale Sandro Pertini, Rome, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Torre, Roma
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), San Donato Milanese (MI)
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda ospedaliero-universitaria Mater Domini, Catanzaro
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Gastroenterology and Endoscopy Unit IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation, Milan
  - Azienda Ospedaliera Universitaria Policlinico de Modena, Modena
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Policlinico Gemelli - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona Medicina Interna, Salerno
  - Ospedale Mauriziano Umberto I, Torino
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia Gastroenterologia, Udine
- Japan (52):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Fujita Health University, Toyoake, Aichi-ken
  - National Hospital Organization Hirosaki National Hospital, Hirosaki, Aomori
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Kitakyushu Municipal Medical Center, Kitakyusyu-shi, Fukoka
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Yukinoseibokai St. Mary's Hospital, Kurume-shi, Fukuoka
  - Hidaka Coloproctology Clinic, Kurume-shi, Fukuoka
  - Gunma University Hosptial, Maebashi, Gunma
  - National Hospital Organization Takasaki General Medical Centar, Takasaki, Gunma
  - NHO Mito Medical Center, Ibaraki-machi, HigaShiibaraki-Gun
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa City Hospital, Asahikawa, Hokkaido
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Aoyama Clinic GI Endoscopy & IBD Center, Kobe, Hyōgo
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Ofuna Central Hospital, Kamakura, Kanagawa
  - Kawasaki Municipal Hospital, Kawasaki, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Sankikai Yokohama Shin midori General Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Mie University Hospital, Tsu, Mie-ken
  - Takagi Clinic - Sendai, Sendai, Miyagi
  - Nagaoka Chuo General Hospital, Nagaoka-shi, Niigata
  - Ishida Clinic of IBD and Gastroenterology, Ōita, Oita Prefecture
  - Sai Gastroenterology, proctology, Fujiidera, Osaka
  - NHO Osaka National Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saga-Ken Medical Center Koseikan, Saga, Saga-ken
  - Kumagaya General Hospital, Kumagaya-shi, Saitama
  - Matsuda Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical And Dental University Medical Hospital, Bunkyō, Tokyo
  - Showa University Koto Toyosu Hospital, Koto-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-Ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - JHCO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Mitsui Memorial Hospital, Chiyoda-ku, Tokyo-To
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo-To
  - Fukuoka University Hospital, Fukuoka
  - Sameshima Hospital, Kagoshima
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Okayama University Hospital, Okayama
  - Infusion Clinic, Osaka
  - Tokitokai Tokito Clinic, Saitama
  - Toyama Prefectural Central Hospital, Toyama
- Latvia (3):
  - Pauls Stradins Clinical Univeristy Hospital, Riga, Rīga
  - Digestive Diseases Center "Gastro", Riga
  - Riga Eastern Clinical University Hospital, Riga
- Lithuania (5):
  - Respublikine Panevezio Ligonine, Panevezys, Panevėžys
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Republic Hospital of Klaipeda, Klaipėda
  - Klaipeda Seamen's Hospital, Klaipėda
  - Vilnius University Hospital Santariskiu Clinics, Vilnius
- Malaysia (5):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Ampang, Ampang, Selangor
- Mexico (7):
  - Clinical Research Institute S C, Tlalnepantla, Edo de Mex
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V., Zapopan, Jalisco
  - Clinicos Asociados BOCM, S.C., Mexico City, Mexico City
  - Centro de Investigación Clínica Acelerada, Mexico City, Mexico City
  - Centro Para el Desarrollo de la Medicina y de Asistencia Med S.C, Culiacán, Sinaloa
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Sociedad de Metabolismo y Corazon, Veracruz
- Netherlands (4):
  - St Elisabeth Ziekenhuis, Tilburg, North Brabant
  - Amsterdam UMC, locatie AMC, Amsterdam, North Holland
  - Bernhoven Ziekenhuis, Uden
  - UMC Utrecht, Dept. of Internal Medicine, MDL, Utrecht
- Poland (24):
  - Szpital Uniwersytecki Nr 2 im. dr J. Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Topolowa Medicenter, Krakow, Lesser Poland Voivodeship
  - Medicenter Nowy Targ, Nowy Targ, Lesser Poland Voivodeship
  - Nzoz Formed, Wadowice, Lesser Poland Voivodeship
  - LexMedica, Wroclaw, Lower Silesian Voivodeship
  - ZOZ Gastromed, Lublin, Lublin Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - NZOZ Vivamed, Warsaw, Masovian Voivodeship
  - Endoskopia sp z o. o, Sopot, Pomeranian Voivodeship
  - SONOMED Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Promedica Dental Clinic, Będzin
  - All-Medicus, Katowice
  - Indywidualna Specjalistyczna Praktyka Lekarska, Knurów
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Gastromed Kopoń Zmudziński I Wspólnicy Spółka Jawna Specjalistyczne Centrum Gastrologii I Endoskopii, Torun
  - Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Zdrowia MDM, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - PlanetMed Sp.z o.o., Wroclaw
  - ETG Zamosc, Zamość
  - KO-Med Centrum Medyczne, Staszów, Świętokrzyskie Voivodeship
- Romania (7):
  - CCBR Clinical Research, Bucharest, București
  - MedLife Grivita, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Hifu Terramed Conformal SRL, Bucharest
  - Centrul Medical Unirea SRL, Bucharest
  - Spital Pelican Oradea, Oradea
- Russia (30):
  - Scientific Centre of Reconstructive and Restorative Surgery, Irkutsk, Irkutsk Oblast
  - Karelia Republican Hospital V.A. Baranova, Petrozavodsk, Kareliya, Respublika
  - Nizhny Novgorod Regional Hospital N.A. Semashko, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Private Healthcare Institution Clinical Hospital Russian Railways - Medicine of Nizhniy Novgorod, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Novosibirsk GastroCenter, Novosibirsk, Novosibirsk Oblast
  - Rostov State Medical University, Rostov-on-Don, Rostov Oblast
  - Scientific research center ECO-security, Saint Petersburg, Sankt-Peterburg
  - Multidisciplinary Medical Clinic "Anthurium", Barnaul
  - Medical and Sanitary Division of Severstal, Cherepovets
  - Alliance Biomedical URAL Group, Izhevsk
  - Clinical Trials Center of Medical Institute, Kaliningrad
  - State Autonomous Institution of Healthcare "Republican Clinical Hospital of the Ministry of Healthcare of Republic Tatarstan", Kazan'
  - SIH Kemerovo Regional Clinical Hosptial, Kemerovo
  - SBHI Regional Clinical Hospital #2 MoH of Krasnodar region, Krasnodar
  - Medical rehabilitation center, Moscow
  - LLC "Medicine Center SibNovoMed", Novosibirsk
  - Clinical Diagnostic Center Ultramed, Omsk
  - City Mariinskaya Hospital, Saint Petersburg
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Saint-Petersburg City Hospital of Saint Elizabeth, Saint Petersburg
  - Non-state Healthcare Institution "Roadway Clinical Hospital of OJSC Russian Railways", Saint Petersburg
  - Saint Petersburg State Medical University n.a. Pavlov I.P., Saint Petersburg
  - LLC Gastroenterology Centre Expert, Saint Petersburg
  - SBIH City Clinical Hospital #31, Saint Petersburg
  - OOO "OrKli", Saint Petersburg
  - Medical Institute REAVIZ, Samara
  - Stavropol State Medical Academy, Stavropol
  - SBI of Healthcare of Leningrad region "Clinical Interregional Hospital of Tosno, Tosno
  - Yaroslavl Municipal HI Clinical Hospital #8, Yaroslavl
  - LLC MA New Hospital, Yekaterinburg
- Serbia (9):
  - Zemun Medical Centre, Zemun, Beograd
  - University Medical Center "Bezanijska kosa", Belgrade, NAP
  - Regional Hospital Dr Radivoj Simonovic Sombor, Sombor, Vojvodina
  - Sremska Mitrovica Health Centre, Sremska Mitrovica, Vojvodina
  - General Hospital "Djordje Joanovic", Zrenjanin, Vojvodina
  - Clinical Hospital Center Zvezdara, Belgrade
  - Clinical Center Kragujevac Gastroenterohepatology Clinic, Kragujevac
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital Uzice, Užice
- Slovakia (7):
  - KM Management, Nitra, Nitra Region
  - Gastro, Prešov, Presov
  - Endomed, s.r.o., Vranov N. Toplou, Presov
  - Alian, s.r.o., Bardejov, Slovak Republic
  - Fakultna nemocnica s poliklinikou Roosevelta Banska Bystrica, Banská Bystrica
  - Univerzitna nemocnica Bratislava-Nemocnica Stare Mesteo, Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
- South Korea (11):
  - Severance Hospital, Yonsei University Health System, Wŏnju, Gangwon-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul, Korea
  - Asan Medical Center, Seoul, Korea
  - Dong-A University Hospital, Busan, Pusan-Kwangyǒkshi
  - Kangbuk Samsung Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon, Taejǒn-Kwangyǒkshi
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Medical Center Chilgok Hospital, Daegu
  - Yeungnam Univeristy Medical Center, Daegu
- Spain (14):
  - Hospital Universitario Virgen Del Rocio, Seville, Andalusia
  - Hospital Universitari Son Espases, Palma de Mallorca, Baleares Islands
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital De Fuenlabrada, Fuenlabrada, Madrid
  - Complejo Hospitalario De Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de Sagunto y C.E., Sagunto, Valencia
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Instituto de Ciencias Médicas, Alicante
  - Hospital Universitario Reina Sofia Comite Etico, Córdoba
  - Hospital Universitari de Girona, Girona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario La Paz, Madrid
- Switzerland (4):
  - Inselspital Bern, Bern
  - Gastroenterologische Praxis Balsiger, Seibold & Partner, Bern
  - Kantonsspital St.Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - Health management center, Taipei
- Turkey (Türkiye) (7):
  - Gazi University Faculty of Medicine, Beşevler, Ankara
  - Hacettepe University Faculty of Medicine, Sihhiye, Ankara
  - Antalya Egitim ve Arastırma Hastanesi, Kocaeli, Antayla
  - Acibadem Universitesi - Acibadem Kozyatagi Hastanesi, Kadıköy, Istanbul
  - Kocaeli University Medical Faculty Hospital, İzmit, Kocaeli
  - Mersin University Medical Faculty, Yenişehir, Mersin
  - Ege Universitesi Hastanesi, Izmir
- Ukraine (23):
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - City Clinical Hospital #2, Kharkiv, Kharkivs’ka Oblast’
  - Kherson City Clinical Hospital, Kherson, Kherson Oblast
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kiev, Kyiv Oblast
  - Lviv Railway Clinical Hospital, Lviv, Lviv Oblast
  - Lviv Regional Endocrinology Dispensary, Lviv, Lviv Oblast
  - Municipal non-profit enterprise "Lviv Territorial Medical Union "Multidisciplinary Clinical Hospital of Em -T, Lviv, Lviv Oblast
  - Poltova Oblast Clinical Hospital IM.M.V.Sklifosovskoho, Poltava, Poltava Oblast
  - Diaservis - Medical and Diagnostic Center, Zaporizhzhia, Zaporizhzhia Oblast
  - Medical Center of Limited Liability Company Medical Center Clinic of Family Medicine, Dnipro
  - Kharkiv City Student Hospital, Kharkiv
  - GI L.T. Malaya TI Namsu, Kharkiv
  - Treatment-Diagnostic Center of Private Enterprise of PPC Atsynus, Kropyvnytskyi
  - Kyiv Municipal Clinical Hospital #1, Kyiv
  - Communal institution of the Kyiv Regional Council "Kyiv Regional Clinical Oncology Dispensary", Kyiv
  - Communal Enterprise "Odesa Regional Clinical Hospital", Odesa
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Vinnytsia RCH of Veterans of War Dept of Therapy#1 Vinnytsia M.I.Pyrogov NMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - M.I. Pyrogov Regional Clinical Hospital, Vinnytsia
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - Private Small Enterprise, Medical Center Pulse, Vinnytsia
  - Communal Institution of Kyiv Regional Council Kyiv Regional Hospital #2, Zaporizhzhia
- United Kingdom (9):
  - Queens Hospital, Romford, Essex
  - Fairfield General Hospital, Bury, Great Britain
  - Royal Hampshire County Hospital, Winchester, Hants
  - St Thomas' Hospital, Great Maze Pond, London
  - Ninewells Hospital, Dundee, Scotland
  - Whipps Cross University Hospital, London, Surrey
  - Morriston Hospital, Swansea, Swansea [Abertawe Gb-ata]
  - St James's University Hospital, Leeds, Vinnytsia
  - Queen Elizabeth University Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Clemow DB, Dubinsky MC, Baygani SK, Sands BE, Keohane A, Danese S, Schreiber S, Walsh AJ, Hibi T, Gibble TH, Moses RE, Travis SPL. Bowel urgency in ulcerative colitis: effect of baseline urgency and change in urgency in response to mirikizumab. J Patient Rep Outcomes. 2025 Jul 1;9(1):75. doi: 10.1186/s41687-025-00906-0. PMID 40591171
- [Derived] Panaccione R, Chan-Diehl F, Baygani S, Fisher DA, Moses RE, Siegmund B, Walsh A, Kobayashi T, Dulai PS, Travis S. Fecal Calprotectin and C-Reactive Protein Association With Histologic and Endoscopic Endpoints in Mirikizumab-Treated Patients With Ulcerative Colitis. Crohns Colitis 360. 2025 Jun 14;7(2):otaf043. doi: 10.1093/crocol/otaf043. eCollection 2025 Apr. PMID 40589947
- [Derived] Sands BE, D'Haens G, Clemow DB, Irving PM, Johns JT, Gibble TH, Abreu MT, Lee SD, Hisamatsu T, Kobayashi T, Dubinsky MC, Vermeire S, Siegel CA, Peyrin-Biroulet L, Moses RE, Milata J, Panaccione R, Dignass A. Three-Year Efficacy and Safety of Mirikizumab Following 152 Weeks of Continuous Treatment for Ulcerative Colitis: Results From the LUCENT-3 Open-Label Extension Study. Inflamm Bowel Dis. 2025 Jul 7;31(7):1876-1890. doi: 10.1093/ibd/izae253. PMID 39448057
- [Derived] Danese S, Dignass A, Matsuoka K, Ferrante M, Long M, Redondo I, Moses R, Maier S, Hunter Gibble T, Morris N, Milch C, Abreu MT. Early and Sustained Symptom Control with Mirikizumab in Patients with Ulcerative Colitis in the Phase 3 LUCENT Programme. J Crohns Colitis. 2024 Nov 4;18(11):1845-1856. doi: 10.1093/ecco-jcc/jjae088. PMID 38869019
- [Derived] Long MD, Schreiber S, Hibi T, Gibble TH, Fisher DA, Park G, Moses RE, Higgins PDR, Lindsay JO, Lee SD, Escobar R, Jairath V. Association of Bowel Urgency With Quality-of-Life Measures in Patients With Moderately-to-Severely Active Ulcerative Colitis: Results From Phase 3 LUCENT-1 (Induction) and LUCENT-2 (Maintenance) Studies. Crohns Colitis 360. 2024 Jan 6;6(1):otae001. doi: 10.1093/crocol/otae001. eCollection 2024 Jan. PMID 38313767
- [Derived] Sands BE, Feagan BG, Hunter Gibble T, Traxler KA, Morris N, Eastman WJ, Schreiber S, Jairath V, Long MD, Armuzzi A. Mirikizumab Improves Quality of Life in Patients With Moderately-to-Severely Active Ulcerative Colitis: Results From the Phase 3 LUCENT-1 Induction and LUCENT-2 Maintenance Studies. Crohns Colitis 360. 2023 Nov 7;5(4):otad070. doi: 10.1093/crocol/otad070. eCollection 2023 Oct. PMID 38034882
- [Derived] Chua L, Friedrich S, Zhang XC. Mirikizumab Pharmacokinetics in Patients with Moderately to Severely Active Ulcerative Colitis: Results from Phase III LUCENT Studies. Clin Pharmacokinet. 2023 Oct;62(10):1479-1491. doi: 10.1007/s40262-023-01281-z. Epub 2023 Aug 23. PMID 37610533
- [Derived] D'Haens G, Dubinsky M, Kobayashi T, Irving PM, Howaldt S, Pokrotnieks J, Krueger K, Laskowski J, Li X, Lissoos T, Milata J, Morris N, Arora V, Milch C, Sandborn W, Sands BE; LUCENT Study Group. Mirikizumab as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2023 Jun 29;388(26):2444-2455. doi: 10.1056/NEJMoa2207940. PMID 37379135
- [Derived] Magro F, Pai RK, Kobayashi T, Jairath V, Rieder F, Redondo I, Lissoos T, Morris N, Shan M, Park M, Peyrin-Biroulet L. Resolving Histological Inflammation in Ulcerative Colitis With Mirikizumab in the LUCENT Induction and Maintenance Trial Programmes. J Crohns Colitis. 2023 Oct 20;17(9):1457-1470. doi: 10.1093/ecco-jcc/jjad050. PMID 37057827
- See also: An Induction Study of Mirikizumab in Participants With Moderately to Severely Active Ulcerative Colitis (LUCENT 1) — https://trials.lillytrialguide.com/en-US/trial/282m4A1tIAKOegkOgG02mg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Main study: Participants were randomized in a 3:1 ratio to 300 milligrams (mg) of mirikizumab intravenously (IV) every 4 weeks (Q4W) or placebo IV Q4W.
  China Maximized Extended Enrollment (ME2): This is an extension phase of the main study, with an additional 166 participants enrolled in China. Safety was monitored and data was reported under Adverse Events (AE) section.
Pre-assignment Details: As pre-specified in the analysis plan, outcome measures were not reported for the Maximum Extended Enrollment (ME2) arms/groups, as no formal efficacy analysis was pre-specified for the ME2 cohorts but only for the main global study arms/groups
Groups:
- Placebo IV Q4W; Placebo IV Q4W ME2 Cohort: Placebo given as an IV infusion Q4W on Weeks 0, 4, 8 for 12 weeks.
- 300 mg Mirikizumab IV Q4W; 300 mg Mirikizumab IV Q4W ME2 Cohort: 300 mg mirikizumab given as an IV infusion Q4W on Weeks 0, 4, 8 for 12 weeks.
Period: Overall Study
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W | Placebo IV Q4W ME2 Cohort | 300 mg Mirikizumab IV Q4W ME2 Cohort
Started | 322 | 959 | 41 | 125
Received at Least One Dose of Study Drug | 321 | 958 | 41 | 125
Completed | 285 | 920 | 36 | 116
Not Completed | 37 | 39 | 5 | 9
Not completed — Adverse Event | 23 | 15 | 3 | 2
Not completed — Withdrawal by Subject | 8 | 5 | 1 | 0
Not completed — Lack of Efficacy | 5 | 5 | 0 | 2
Not completed — Protocol Violation | 1 | 5 | 1 | 3
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0
Not completed — Insufficient Diary Data | 0 | 2 | 0 | 0
Not completed — Non- compliance to Protocol | 0 | 1 | 0 | 0
Not completed — COVID-19 Related Study Disruption | 0 | 2 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W | Placebo IV Q4W ME2 Cohort | 300 mg Mirikizumab IV Q4W ME2 Cohort | Total
Number analyzed (Participants) | 322 | 959 | 41 | 125 | 1447
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (13.78) | 42.8 (13.83) | 49.4 (15.43) | 44.0 (13.88) | 42.8 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 367 | 13 | 46 | 566
  Male | 182 | 592 | 28 | 79 | 881
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 22 | 0 | 0 | 31
  Not Hispanic or Latino | 27 | 92 | 25 | 84 | 228
  Unknown or Not Reported | 286 | 845 | 16 | 41 | 1188
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 10 | 0 | 0 | 12
  Asian | 68 | 224 | 41 | 125 | 458
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 10 | 0 | 0 | 12
  White | 247 | 704 | 0 | 0 | 951
  More than one race | 2 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 9 | 0 | 0 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 3 | 8 | 0 | 0 | 11
  Australia | 4 | 10 | 0 | 0 | 14
  Austria | 2 | 6 | 0 | 0 | 8
  Belgium | 3 | 6 | 0 | 0 | 9
  Canada | 11 | 23 | 0 | 0 | 34
  China | 2 | 16 | 41 | 125 | 184
  Croatia | 1 | 1 | 0 | 0 | 2
  Czechia | 20 | 35 | 0 | 0 | 55
  Denmark | 0 | 7 | 0 | 0 | 7
  France | 15 | 49 | 0 | 0 | 64
  Germany | 6 | 33 | 0 | 0 | 39
  Hungary | 7 | 16 | 0 | 0 | 23
  India | 21 | 62 | 0 | 0 | 83
  Ireland | 0 | 1 | 0 | 0 | 1
  Israel | 3 | 14 | 0 | 0 | 17
  Italy | 12 | 25 | 0 | 0 | 37
  Japan | 35 | 102 | 0 | 0 | 137
  Latvia | 6 | 24 | 0 | 0 | 30
  Lithuania | 6 | 16 | 0 | 0 | 22
  Malaysia | 0 | 6 | 0 | 0 | 6
  Mexico | 2 | 10 | 0 | 0 | 12
  Netherlands | 2 | 9 | 0 | 0 | 11
  Poland | 32 | 104 | 0 | 0 | 136
  Romania | 2 | 13 | 0 | 0 | 15
  Russia | 28 | 79 | 0 | 0 | 107
  Serbia | 8 | 13 | 0 | 0 | 21
  Slovakia | 3 | 21 | 0 | 0 | 24
  South Korea | 5 | 23 | 0 | 0 | 28
  Spain | 7 | 15 | 0 | 0 | 22
  Switzerland | 2 | 9 | 0 | 0 | 11
  Taiwan | 0 | 3 | 0 | 0 | 3
  Turkey | 5 | 6 | 0 | 0 | 11
  Ukraine | 26 | 68 | 0 | 0 | 94
  United Kingdom | 7 | 11 | 0 | 0 | 18
  United States | 36 | 115 | 0 | 0 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission at Week 12
Description: Clinical remission at week 12 is defined as achieving a modified Mayo score (MMS) subscore for rectal bleeding=0, stool frequency=0 or 1 with ≥ 1 point decrease from baseline, and endoscopy=0 or 1 (excluding friability), excluding consideration of Physician's Global Assessment (PGA).
  Stool frequency subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal); Rectal bleeding subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed); Endoscopy subscore, based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The confidence interval of 99.88% was chosen to match the significance level.
Time Frame: Week 12
Population: Modified Intention-to-treat population (mITT): All randomized participants who received at least one dose of study drug and who had the modified Mayo score measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
  As pre-specified in the analysis plan, outcome measures were not reported for ME2 arms,as no formal efficacy analysis was pre-specified for ME2 cohort but only for the main global study arms/groups.
Measure: Number (99.88% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
percentage of participants | 13.3 [6.9 to 19.6] | 24.2 [19.5 to 28.9]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.00006, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.1, 99.875% CI 2-sided [3.2 to 19.1]

2. Secondary Outcome: Percentage of Participants With Clinical Response at Week 12
Description: Clinical response at week 12 is defined as a decrease in the 9-point modified Mayo score (MMS) [rectal bleeding, stool frequency and the endoscopic findings] inclusive of >= 2 points and >=30% from baseline with either a decrease of rectal bleeding subscore of >=1 or rectal bleeding subscore of 0 or 1.The MMS is a composite score of ulcerative colitis disease activity calculated as the sum of three subscores: Stool frequency subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal); Rectal bleeding subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed); Endoscopy subscore, based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding,ulceration).The MMS ranges from 0 to 9 points,with higher scores representing more severe disease. The confidence interval of 99.88% was chosen to match the significance level.
Time Frame: Week 12
Population: mITT Population: All randomized participants who received at least one dose of study drug and who had the modified Mayo score measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
  As pre-specified in the analysis plan, outcome measures were not reported for ME2 arms,as no formal efficacy analysis was pre-specified for ME2 cohort but only for the main global study arms/groups.
Measure: Number (99.88% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
percentage of participants | 42.2 [32.9 to 51.5] | 63.5 [58.2 to 68.8]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.4, 99.875% CI 2-sided [10.8 to 32.0]

3. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission at week 12 is defined as achieving a Mayo endoscopic subscore of 0 or 1 (excluding friability) at Week 12. Endoscopy subscore is based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration);
  The Mayo endoscopic score ranges from 0 to 3 points, with higher scores representing more severe disease.
  The confidence interval of 99.88% was chosen to match the significance level.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (99.88% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
percentage of participants | 21.1 [13.4 to 28.8] | 36.3 [31.0 to 41.6]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.4, 99.875% CI 2-sided [6.3 to 24.5]

4. Secondary Outcome: Percentage of Participants With Symptomatic Remission at Week 12
Description: Symptomatic remission at week 12 is defined as a Mayo subscore for rectal bleeding=0, stool frequency=0 or 1 with ≥ 1 point decrease from baseline.
  Stool frequency subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal).
  Rectal bleeding subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed).
  The confidence interval of 99.88% was chosen to match the significance level.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (99.88% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
percentage of participants | 27.9 [22.8 to 33.0] | 45.5 [42.2 to 48.8]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.5, 99.875% CI 2-sided [11.4 to 23.6]

5. Secondary Outcome: Percentage of Participants With Symptomatic Response at Week 12
Description: Symptomatic response at week 12 is defined as ≥30% decrease from baseline in the sum of stool frequency and rectal bleeding subscores.
  Stool frequency subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal).
  Rectal bleeding subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed). The sum of stool frequency and rectal bleeding subscores ranges from 0 to 6.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
percentage of participants | 52.4 [46.7 to 58.1] | 72.0 [69.0 to 75.0]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.2, 95% CI 2-sided [13.8 to 26.6]

6. Secondary Outcome: Percentage of Participants With Histologic Remission at Week 12
Description: Histologic remission was assessed using the Geboes histologic scoring system developed for assessment of histologic disease activity in ulcerative colitis. Remission was defined as Geboes histological subscore of 0 for grades: 2b (lamina propria neutrophils), and 3 (neutrophils in epithelium), and 4 (crypt destruction), and 5 (erosion or ulceration).
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
percentage of participants | 15.6 [11.5 to 19.8] | 29.3 [26.2 to 32.3]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.7, 95% CI 2-sided [8.6 to 18.7]

7. Secondary Outcome: Percentage of Participants With Endoscopic Response at Week 12
Description: Endoscopic response at week 12 is defined as achieving at least a 1 point decrease from baseline in the Mayo endoscopic subscore.
  The Mayo endoscopic subscore ranges from 0 to 3 points, with higher scores representing more severe disease.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
percentage of participants | 36.1 [30.6 to 41.5] | 55.4 [52.1 to 58.7]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.00001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.5, 95% CI 2-sided [13.2 to 25.8]

8. Secondary Outcome: Change From Baseline to Week 12 in Bowel Urgency Based on the Urgency Numeric Rating Scale (NRS)
Description: The Urgency NRS is a single participant reported item that measures the severity for the urgency (sudden or immediate need) to have a bowel movement in the past 24 hours using an 11-point NRS ranging from 0 (no urgency) to 10 (worst possible urgency).Higher scores indicate more severe urgency. Least square (LS) Mean was calculated using mixed model repeated measures (MMRM) model for post-baseline measures: The MMRM model includes: treatment, baseline value, visit, interaction of baseline value-by-visit, interaction of treatment-by-visit, prior biologic or tofacitinib failure (yes/no), baseline corticosteroid use (yes/no), baseline disease activity (MMS: [4-6] or [7-9]), and region (North America/Europe/Other).
Time Frame: Baseline, Week 12
Population: mITT population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least one post-baseline urgency NRS measurement. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
  As pre-specified in the analysis plan, outcome measures were not reported for ME2 arms,as no formal efficacy analysis was pre-specified for ME2 cohort but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
score on a scale | -1.63 (0.141) | -2.59 (0.083)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.00001, Mixed Models Analysis; Mean Difference (Net) = -0.95, 99.875% CI 2-sided [-1.47 to -0.44], Standard Error of Mean 0.159 — The confidence interval of 99.875 % was chosen to match the significance level

9. Secondary Outcome: Change From Baseline to Week 12 in Health Related Quality of Life: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score
Description: The IBDQ is a 32-item participant-completed questionnaire that measures 4 aspects of subjects' lives: symptoms directly related to the primary bowel disturbance, systemic symptoms, emotional function, and social function (Guyatt et al. 1989). Responses are graded on a 7-point. Likert scale in which 7 denotes "not a problem at all" and 1 denotes "a very severe problem." Scores range from 32 to 224; a higher score indicates a better quality of life. Least square (LS) Mean was calculated using analysis of covariance (ANCOVA) model for post-baseline measures: The ANCOVA model includes: treatment, baseline value, prior biologic or tofacitinib failure (yes/no), baseline corticosteroid use (yes/no), baseline disease activity (MMS: [4-6] or [7-9]), and region (North America/Europe/Other).
Time Frame: Baseline, Week 12
Population: mITT population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least one post-baseline IBDQ measurement. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
  As pre-specified in the analysis plan, outcome measures were not reported for ME2 arms,as no formal efficacy analysis was pre-specified for ME2 cohort but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 294 | 868
score on a scale | 25.21 (1.798) | 38.42 (1.108)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 13.21, 95% CI 2-sided [9.28 to 17.15], Standard Error of Mean 2.005

10. Secondary Outcome: Change From Baseline to Week 12 in Fecal Calprotectin
Description: Fecal calprotectin is an indicator of inflammation in the colon with higher levels indicative of higher levels of inflammation. Least square (LS) Mean was calculated using mixed model repeated measures (MMRM) model for post-baseline measures: The MMRM model includes: treatment, baseline value, visit, interaction of baseline value-by-visit, interaction of treatment-by-visit, prior biologic or tofacitinib failure (yes/no), baseline corticosteroid use (yes/no), baseline disease activity (MMS: [4-6] or [7-9]), and region (North America/Europe/Other).
Time Frame: Baseline, Week 12
Population: mITT population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least one post-baseline fecal calprotectin measurement. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
  As pre-specified in the analysis plan, outcome measures were not reported for ME2 arms,as no formal efficacy analysis was pre-specified for ME2 cohort but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: milligram per kilogram (mg/kg)
Arm/Group | Placebo IV Q4W | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 206 | 665
milligram per kilogram (mg/kg) | -939.69 (196.557) | -1875.29 (116.138)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 300 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -935.60, 95% CI 2-sided [-1363.64 to -507.55], Standard Error of Mean 218.090

11. Secondary Outcome: Pharmacokinetics (PK): Clearance of Mirikizumab
Description: Clearance of mirikizumab was evaluated. Clearance is estimated based on concentration data collected in the time frame of 0-12 weeks.
Time Frame: Predose on week 0, week 4, week 8 and post dose on week 0, 4 and 12
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
  As pre-specified in the analysis plan, outcome measures were not reported for ME2 arms,as no formal efficacy analysis was pre-specified for ME2 cohort but only for the main global study arms/groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour (L/h)
Arm/Group | 300 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 952
Liters per Hour (L/h) | 0.0224 (38)

ADVERSE EVENTS:
Time Frame: Baseline Up to week 32
Description: All randomized participants who received at least one dose of study drug. MedDRA 24.0 was used for the main global study arms/groups, and MedDRA 26.1 was used for the ME2 arms/groups.
Groups:
- 300 Mirikizumab IV Q4W; 300 mg Mirikizumab IV Q4W ME2 Cohort: 300 mg mirikizumab given as an IV infusion Q4W on Weeks 0, 4, 8 for 12 weeks.
Arm/Group | Placebo IV Q4W | 300 Mirikizumab IV Q4W | Placebo IV Q4W ME2 Cohort | 300 mg Mirikizumab IV Q4W ME2 Cohort
All-Cause Mortality (participants affected / at risk) | 0/321 | 0/958 | 0/41 | 0/125
Serious Adverse Events (participants affected / at risk) | 17/321 | 27/958 | 7/41 | 10/125
Other Adverse Events (participants affected / at risk) | 18/321 | 31/958 | 11/41 | 25/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV Q4W (N=321) | 300 Mirikizumab IV Q4W (N=958) | Placebo IV Q4W ME2 Cohort (N=41) | 300 mg Mirikizumab IV Q4W ME2 Cohort (N=125)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 10 (10) | 8 (8) | 4 (4) | 4 (4)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile vein thrombosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV Q4W (N=321) | 300 Mirikizumab IV Q4W (N=958) | Placebo IV Q4W ME2 Cohort (N=41) | 300 mg Mirikizumab IV Q4W ME2 Cohort (N=125)
Anaemia (Blood and lymphatic system disorders) | 18 (18) | 31 (32) | 4 (4) | 8 (8)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol: AMAN 05 Protocol (a)_Redacted (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03518086/Prot_000.pdf
  • Study Protocol: AMAN 05 ME2 Protocol Addenda (5)_Redacted (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03518086/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03518086/SAP_002.pdf
  • Statistical Analysis Plan: I6T-MC-AMAN ME2 Statistical Analysis Plan Addendum Version 1 (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT03518086/SAP_003.pdf